CLINICAL TRIAL: NCT06135896
Title: An Open-label, Randomized, Multicenter, Phase II Tripegfilgrastim Trial to Reduce the Risk of Severe Neutropenia in Patients With Unresectable Pancreaticobiliary Cancers
Brief Title: Tripegfilgrastim Trial to Reduce the Risk of Severe Neutropenia in Patients With Unresectable Pancreaticobiliary Cancers
Acronym: Dulastin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Myung Woo, medical doctor, Senior scientist, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCC2023-0235
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Pancreatic Cancer; Unresectable Bile Duct Carcinoma; Unresectable Biliary Tract Carcinoma
Keywords: Unresectable Pancreatic Cancer; Unresectable Bile Duct Carcinoma; Unresectable Biliary Tract Carcinoma

STUDY DESIGN:
Intervention Model Description: * Clinical trial phase: Phase 2
  * Group allocation: Randomized controlled trial
  * Research perspective: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): * Premedication: depending on the center (Ondansetron 8 mg +Dextrose 5% 50 mL, MIV, Dexamethason 10 mg IV, and Atropine sulfate 0.25 mg [0.5 amp] SC)
  * Onivyde 70 mg/m2 + Dextrose 5% 500 mL (bag), and MIV for 90 min
  * Leucovorin 400 mg/m2 + Dextrose 5% 500 mL (bag), and MIV for 30 min
  * 5-FU (2400 mg/m2) + Dextrose 5% 500 mL (bag) and MIV for 46 h
  * Tripegfilgrastim 6 mg SC administered 24 h after completing 5-FU infusion The above chemotherapy will be administered every two weeks
  Interventions: Drug: Tripegfilgrastim
- Control Group (No Intervention): * Premedication: depending on center (Ondansetron 8 mg+Dextrose 5% 50 mL, MIV, Dexamethason 10 mg IV, and Atropine sulfate 0.25 mg [0.5 amp] SC)
  * Onivyde 70 mg/m2 + Dextrose 5% 500 mL (bag), and MIV for 90 min
  * Leucovorin 400 mg/m2 + Dextrose 5% 500 mL (bag), and MIV for 30 min
  * 5-FU (2400 mg/m2) + Dextrose 5% 500 mL (bag), and MIV for 46 h The following medication will be provided in the event that the patient develops febrile neutropenia after the above chemotherapy
  * Tripegfilgrastim 6 mg SC administered 24 h after stopping 5-FU. In the event of neutropenia, chemotherapy will be paused until the patient recovers, and then restarted after recovery.
  * The above chemotherapy will be administered every two weeks.

INTERVENTIONS:
Drug: Tripegfilgrastim — Tripegfilgrastim to reduce the risk of severe neutropenia in patients with unresectable pancreaticobiliary cancers
  Other Names: Dulastin
  Arms: Treatment Group

SUMMARY:
* Clinical trial phase: Phase 2
* Intervention model: Control group
* Group allocation: Randomized controlled trial
* Research perspective: Prospective study
* Participating centers: Multicenter study
* Definition of the intervention period: Based on the RECIST 1.1 guidelines, patients will receive treatment until dropout due to disease progression or unacceptable toxicity related to the trial drug. Patients will be followed up with to assess survival every 2 months until either death or the end of the trial, whichever is first.
* The intervention period is from the date of IRB approval to December 31st, 2025
* The follow-up duration is one year, and the statistical analysis duration is six months
* The total research period is from the date of IRB approval to June 30th, 2026

DETAILED DESCRIPTION:
Pancreatic cancer and Bile duct cancer are the 8th and 9th leading causes of all cancer in Korea, have 5-year survival rates of approximately 20%, and unresectable cancers show a poor prognosis of approximately 5%. The first-line treatment recommended for unresectable pancreaticobiliary cancer is chemotherapy. FOLFIRINOX or gemcitabine/nab-paclitaxel combination therapy is recommended for pancreatic cancer, and gemcitabine/cisplatin combination therapy is recommended for bile duct cancer. Recently, anticancer therapy advances have led to an increase in survival for pancreaticobiliary cancer patients, and more than half of patients receive secondary chemotherapy due to disease progression after first-line treatment. Recently, with the introduction of nanoliposomal irinotecan (nal-IRI) and the clinical outcomes of Phase 3 NAPOL-1 trial and the Phase 2b NIFTY trial, nal-IRI/5-FU/LV combination therapy is being used as second-line chemotherapy following gemcitabine treatment. Granulocyte colony-stimulating factors (G-CSFs) (filgrastim, pegfilgrastim, and tripegfilgrastim) can be used for neutropenia prevention and treatment. In particular, pegylated G-CSF can reduce patient discomfort due to its long retention time. In a retrospective study analyzing the use of G-CSF for primary neutropenia prevention in Korea, pancreatic cancer patients who received FOLFIRINOX treatment that exhibited neutropenia and FN were significantly reduced from 55.6% to 31.6% (P = 0.003) and from 18.5% to 1.8% (P = 0.002), respectively. Similarly, in a retrospective study in Japan, preventive pegylated G-CSF treatment reduced the incidence of FN from 23% to 0%, and in a double-blinded, randomized, phase 3 breast cancer clinical trial, pegylated G-CSF treatment significantly reduced the incidence of FN from 68.8% to 1.2%. In a retrospective study of non-small cell lung cancer, another solid cancer, the incidence of FN in the preventive pegylated G-CSF treatment group was 0%, compared to an incidence of 50% in the control group.

However, no studies have evaluated the efficacy of G-CSF in pancreaticobiliary cancer patients receiving nal-IRI/5-FU/LV combination therapy yet. Hence, our objective was to report the effects of pegylated G-CSF on preventing severe neutropenia in patients receiving nal-IRI/5-FU/LV combination chemotherapy for unresectable pancreaticobiliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 19 years old, diagnosed with unresectable pancreaticobiliary cancer, and scheduled to receive chemotherapy using nal-IRI/5-FU/LV combination chemotherapy

Exclusion Criteria:

* Patients who refuse to sign the consent form Patients who have previously experienced severe neutropenia during chemotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | through study completion, an average of 1 year
  Severe neutropenia incidence

SECONDARY OUTCOMES:
neutropenia incidence | through study completion, an average of 1 year
  All grades of neutropenia incidence
Febrile neutropenia | through study completion, an average of 1 year
  Febrile neutropenia incidence
emergency department visits | through study completion, an average of 1 year
  Frequency of unexpected emergency department visits and length of stay
Overall survival | through study completion, an average of 1 year
  Overall survival
Progression-free survival | through study completion, an average of 1 year
  Progression-free survival
biomarkers | through study completion, an average of 1 year
  Predictive biomarkers for treatment response analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sangmyung Woo, M.D, Principal Investigator — National Cancer Center
Locations (1):
- NATIONAL CANCER CENTER 323, Ilsan-ro, Ilsandong-gu,, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang MJ, Lim J, Han SS, Park HM, Kim SW, Lee WJ, Woo SM, Kim TH, Won YJ, Park SJ. Distinct prognosis of biliary tract cancer according to tumor location, stage, and treatment: a population-based study. Sci Rep. 2022 Jun 17;12(1):10206. doi: 10.1038/s41598-022-13605-3. PMID 35715440
- [Result] Canton C, Boussari O, Boulin M, Le Malicot K, Taieb J, Dahan L, Lopez A, Lepage C, Bachet JB. Impact of G-CSF Prophylaxis on Chemotherapy Dose-Intensity, Link Between Dose-Intensity and Survival in Patients with Metastatic Pancreatic Adenocarcinoma. Oncologist. 2022 Jul 5;27(7):e571-e579. doi: 10.1093/oncolo/oyac055. PMID 35289915
- [Result] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Result] Yoo C, Im HS, Kim KP, Oh DY, Lee KH, Chon HJ, Kim JH, Kang M, Kim I, Lee GJ, Oh SY, Choi Y, Choi HJ, Kim ST, Park JO, Ryoo BY. Real-world efficacy and safety of liposomal irinotecan plus fluorouracil/leucovorin in patients with metastatic pancreatic adenocarcinoma: a study by the Korean Cancer Study Group. Ther Adv Med Oncol. 2019 Aug 23;11:1758835919871126. doi: 10.1177/1758835919871126. eCollection 2019. PMID 31489036
- [Result] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Result] Yoo C, Kim KP, Jeong JH, Kim I, Kang MJ, Cheon J, Kang BW, Ryu H, Lee JS, Kim KW, Abou-Alfa GK, Ryoo BY. Liposomal irinotecan plus fluorouracil and leucovorin versus fluorouracil and leucovorin for metastatic biliary tract cancer after progression on gemcitabine plus cisplatin (NIFTY): a multicentre, open-label, randomised, phase 2b study. Lancet Oncol. 2021 Nov;22(11):1560-1572. doi: 10.1016/S1470-2045(21)00486-1. Epub 2021 Oct 14. PMID 34656226
- [Result] Chun JW, Woo SM, Lee SH, Choi JH, Park N, Kim JS, Cho IR, Paik WH, Lee WJ, Ryu JK, Kim YT. A real-world analysis of nanoliposomal-irinotecan with 5-fluorouracil and folinic acid as third- or later-line therapy in patients with metastatic pancreatic adenocarcinoma. Ther Adv Med Oncol. 2022 Aug 29;14:17588359221119539. doi: 10.1177/17588359221119539. eCollection 2022. PMID 36062047
- [Result] Jung JH, Shin DW, Kim J, Lee JC, Hwang JH. Primary Granulocyte Colony-Stimulating Factor Prophylaxis in Metastatic Pancreatic Cancer Patients Treated with FOLFIRINOX as the First-Line Treatment. Cancers (Basel). 2020 Oct 27;12(11):3137. doi: 10.3390/cancers12113137. PMID 33120908
- [Result] Sasaki M, Ueno H, Mitsunaga S, Ohba A, Hosoi H, Kobayashi S, Ueno M, Terazawa T, Goto M, Inoue D, Namiki S, Sakamoto Y, Kondo S, Morizane C, Ikeda M, Okusaka T. A phase II study of FOLFIRINOX with primary prophylactic pegfilgrastim for chemotherapy-naive Japanese patients with metastatic pancreatic cancer. Int J Clin Oncol. 2021 Nov;26(11):2065-2072. doi: 10.1007/s10147-021-02001-y. Epub 2021 Aug 8. PMID 34368921
- [Result] Kosaka Y, Rai Y, Masuda N, Takano T, Saeki T, Nakamura S, Shimazaki R, Ito Y, Tokuda Y, Tamura K. Phase III placebo-controlled, double-blind, randomized trial of pegfilgrastim to reduce the risk of febrile neutropenia in breast cancer patients receiving docetaxel/cyclophosphamide chemotherapy. Support Care Cancer. 2015 Apr;23(4):1137-43. doi: 10.1007/s00520-014-2597-1. Epub 2015 Jan 10. PMID 25576433
- [Result] Sahai V, Catalano PJ, Zalupski MM, Lubner SJ, Menge MR, Nimeiri HS, Munshi HG, Benson AB 3rd, O'Dwyer PJ. Nab-Paclitaxel and Gemcitabine as First-line Treatment of Advanced or Metastatic Cholangiocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1707-1712. doi: 10.1001/jamaoncol.2018.3277. PMID 30178032
- [Result] Callingham BA. Some aspects of monoamine oxidase pharmacology. Cell Biochem Funct. 1986 Apr;4(2):99-108. doi: 10.1002/cbf.290040204. No abstract available. PMID 3085974
- [Result] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341